CLINICAL TRIAL: NCT06976892
Title: A Phase I/Ib Trial of Idetrexed (Alpha Folate Receptor Targeted Thymidylate Synthase Inhibitor) in Combination With Olaparib (a PARP Inhibitor) at Different Doses in Patients With Ovarian Cancer (IDOL)
Brief Title: Investigating Idetrexed and Olaparib in Patients With Ovarian Cancer
Acronym: IDOL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Algok Bio Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CCR5978; 1008393 (Registry Identifier: Integrated Research Application System (IRAS))
Record Dates: First submitted 2025-04-03; First posted 2025-05-16 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: High Grade Serous Ovarian Cancer
Keywords: Ovarian Cancer; idetrexed; olaparib
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Maximum Tolerated Dose

STUDY DESIGN:
Intervention Model Description: Up to 4 dose levels of Olaparib in combination with Idetrexed will be explored. Dose Escalation will use a flexible TIme To Event Continual Reassessment Method (TITE-CRM) including time-to-toxicity analysis to account for dose-limiting toxicities that may arise outside the initial DLT period (2 cycles). The TITE-CRM was proposed to handle the problem of long trial duration in Phase 1 trials due to late-onset toxicities. By combining a "backfilling" feature with TITE-CRM, the aim is to significantly shorten trial duration while maintaining a good assessment of the Maximum Tolerated Dose and Recommended Phase 2 Dose. The latter will consider not only the DLT outcomes, but also other parameters including activity and patient tolerability, as well as biomarker response during dose expansion. The proposed trial design ensures that the study has the advantages of both speed and efficiency.
  PLEASE NOTE: INTRA-PATIENT DOSE ESCALATION IS NOT PERMITTED ON THIS STUDY.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Experimental): Patients may be assigned one of four dose levels for the combination of idetrexed and Olaparib:
  * Dose Level 2 (starting dose): 9 mg/m2 idetrexed administered intravenously on days 1 and 15 of each cycle; 300 mg Olaparib administered orally twice per day on days 1-7 and 15-21.
  * Dose Level 1: 9 mg/m2 idetrexed administered intravenously on days 1 and 15 of each cycle; 200 mg Olaparib administered orally twice per day on days 1-7 and 15-21.
  * Dose Level -1: 9 mg/m2 idetrexed administered intravenously on days 1 and 15 of each cycle; 150 mg Olaparib administered orally twice per day on days 1-7 and 15-21.
  * Dose Level 3: 12 mg/m2 idetrexed administered intravenously on days 1 and 15 of each cycle; 200 mg Olaparib administered orally twice per day on days 1-7 and 15-21.
  Interventions: Drug: Dose Level 2 (starting dose); Drug: Dose Level 1; Drug: Dose Level -1; Drug: Dose Level 3
- Dose Expansion (Experimental): Only patients expressing high levels of alpha-folate receptor on their tumours will be eligible. The maximum tolerated dose of Olaparib in combination with idetrexed, based on safety and efficacy data from Dose Escalation, will inform the dose carried forward to Dose Expansion.
  Interventions: Drug: Maximum Tolerated Dose

INTERVENTIONS:
Drug: Dose Level 2 (starting dose) — Idetrexed: 9 mg/m2 I.V. (days 1 & 8) Olaparib: 300 mg P.O. (days1-7, 15-21)
  Arms: Dose Escalation
Drug: Dose Level 1 — Idetrexed: 9 mg/m2 I.V. (days 1 & 8) Olaparib: 200 mg P.O. (days1-7, 15-21)
  Arms: Dose Escalation
Drug: Dose Level -1 — Idetrexed: 9 mg/m2 I.V. (days 1 & 8) Olaparib: 150 mg P.O. (days1-7, 15-21)
  Arms: Dose Escalation
Drug: Dose Level 3 — Idetrexed: 12 mg/m2 I.V. (days 1 & 8) Olaparib: 200 mg P.O. (days1-7, 15-21)
  Arms: Dose Escalation
Drug: Maximum Tolerated Dose — MTD of Olaparib in combination with idetrexed established from Dose Escalation
  Arms: Dose Expansion

SUMMARY:
Two drugs called Idetrexed and olaparib are being evaluated. Idetrexed is a type of drug called an "aFR-targeted thymidylate synthase inhibitor". Idetrexed has been designed to selectively target cancer cells that have a protein called folate receptor on the surface of cancer cells. Thymidylate synthase is key to cancer cells for creating new DNA when they multiply. Blocking the action of thymidylate synthase with a drug like Idetrexed may therefore stop cancers from growing by damaging DNA in cancer cells. Olaparib is a type of drug called a "PARP inhibitor". It prevents cells repairing DNA damage. This leads to cells dying. Combining Idetrexed and olaparib should increase the number of cancer cells dying, especially those cells that have a lot of folate receptors. Cancer cells with a high number of folate receptors should be targeted more than normal healthy cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven high grade serous ovarian cancer refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient.
* Measurable (as defined by RECIST v1.1) or evaluable (based on tumour markers) disease.
* Life expectancy of at least 12 weeks.
* World Health Organisation (WHO) performance status of 0-1 (Appendix 1 of Protocol).
* Haematological and biochemical indices within the ranges shown in Protocol section 4.1.1). These measurements must be performed within one week (Day -7 to Day 1) prior to the patient's first dose of IMP.

Normal (no clinically significant abnormalities) 12-lead ECG, QTcF interval <470 ms

* Pulmonary function test FVC of >70%, DLCOc (DLCO corrected for Hb) of >60%.
* 18 years or over.
* Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up.
* For dose expansion patients only, they must have medium to high α-folate receptor expression according to the Ventana FOLR1-2.1 IHC assay.

Exclusion Criteria:

* Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas, Mitomycin-C) and 4 weeks for investigational medicinal products) before treatment.
* Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or certain Grade 1 toxicities, which in the opinion of the Investigator and the DDU should not exclude the patient.
* Patients with new brain metastases. Patients with treated (surgically excised or irradiated) and stable brain metastases are eligible as long as the treatment was at least 4 weeks prior to initiation of study drug and brain MRI within 2 weeks of initiation of study drug is negative for new metastases.
* Patients with pulmonary metastases.
* History of thoracic radiation or other history likely to create pre-existing lung disease
* Presence of significant clinical ascites and/or pleural effusions.
* Female patients of child-bearing potential (or are already pregnant or lactating). However, those patients who have a negative serum or urine pregnancy test before enrolment and agree to use two forms of contraception (one effective form plus a barrier method) [oral, injected or implanted hormonal contraception and condom; intra-uterine device and condom; diaphragm with spermicidal gel and condom] or agree to sexual abstinence (see Protocol Section 16.5 - Appendix 5), effective from signing the consent form, throughout the trial and for six months afterwards are considered eligible.
* Major thoracic or abdominal surgery from which the patient has not yet recovered.
* Patients with sub-acute bowel obstruction.
* Organ transplant patients.
* At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
* Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
* Patients with history of QT prolongation, clinically significant VT, VF, heart block, MI within 1 year, CHF NYHA Class III or IV, unstable angina, angina within 6 months, or other evidence of clinically significant coronary artery disease/
* Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase I/Ib study of Idetrexed and Olaparib. Participation in an observational trial would be acceptable.
* Inability to tolerate Olaparib.
* Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.
* Confirmed, current COVID-19 infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender women
Enrollment: 33 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Propose a recommended dose/schedule for Phase II evaluation of the combination of Idetrexed and Olaparib | End of Cycle 2 (each cycle is 28 days)
  Endpoint: Maximum tolerated dose/ schedule (MTD) of the combination of Idetrexed and Olaparib based on dose-limiting toxicities (DLT) with target acceptable DLT rate of 25%, and the Recommended Phase II dose (RP2D) and schedule (Dose Escalation only).
Assess the safety and toxicity profile of Idetrexed and Olaparib | End of Cycle 6 (each cycle is 28 days)
  Endpoint: determining causality of each adverse event to Idetrexed and Olaparib and grading severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (Dose Escalation and Dose Expansion).
Evaluate the preliminary anti-tumour activity of the combination of Idetrexed and Olaparib in alpha folate receptor overexpressing high grade serous ovarian cancer | Until patient withdraws due to radiological progression, or begins new line of therapy.
  Endpoint: Objective response rate by the occurrence of Best Overall Response (BOR) per RECIST 1.1 criteria (Dose Expansion only).

SECONDARY OUTCOMES:
Evaluate antitumour activity of the combination of Idetrexed and Olaparib | From date of enrolment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Endpoint: Progression Free Survival (PFS).
Evaluate the preliminary anti-tumour activity of the combination of Idetrexed and Olaparib in ovarian cancer irrespective of alpha folate receptor expression status | From date of enrolment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months.
  Objective response rate.
CA125 responses | From date of enrolment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months.
  Measurement of CA125 levels.

OTHER OUTCOMES:
(Tertiary Objective): Retrospective evaluation of response biomarkers | Within four weeks of patient beginning treatment.
  Alpha-folate expression.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Udai Banerji, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (3):
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Royal Marsden Hospital - Drug Development Unit, Sutton, London
  - Velindre Cancer Centre, Cardiff, Wales

IPD SHARING:
Plan to Share IPD: Undecided